CLINICAL TRIAL: NCT01109667
Title: The Effects of Different Reagents on Coagulation Tests: Innovin Versus Thromborel-S.
Brief Title: Differences in Coagulation Test Kits
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas Hospital (Other)
Other Study IDs: EPK-235
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-01

CONDITIONS: Effect of Different Reagents.; Oral Anticoagulant Therapy
Keywords: Thromboplastin, Prothrombin, Diagnostic Reagent Kits, International Normalized Ratio, Laboratory Tests.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- oral anticoagulant: Patients receiving and not receiving oral anticoagulant therapy.
- INR Level: Group I: Patients not receiving OAT, Group II: Patients under OAT and INR values in good therapeutic range and Group III: Patients under OAT and INR values over the therapeutic range.

SUMMARY:
The aim of this study is to assess the effect of Innovin® reagent on laboratory results when compared with the Thromborel® S.

DETAILED DESCRIPTION:
Thromboplastins are the screening tests which are used in the diagnosis of acquired or inherited disorders of the coagulation system but still, alterations between various thromboplastin preparations in the measurements remains a problem.Blood samples are going to drawn from patients receiving and not receiving oral anticoagulant therapy (OAT) during their routine laboratory tests. Samples are subjected to analysis by using Thromborel® S and Innovin® reagents. Mean International Normalized Ratio (INR), prothrombin time and fibrinogen values are going to compared. To further study the importance of this phenomenon the cohort will be divided into three subgroups according to the INR values as Group I: Patients not receiving OAT, Group II: Patients under OAT and INR values in good therapeutic range and Group III: Patients under OAT and INR values over the therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

Routine control patients receiving and not receiving oral anticoagulant therapy

Exclusion Criteria:

Hemolytic and/or lipemic samples were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving and not receiving oral anticoagulant therapy
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Turkiye Yuksek Ihtisas Hospital, Ankara, Turkey (Türkiye)